CLINICAL TRIAL: NCT02056483
Title: Optimized Rehabilitation: A Randomized Study of Systematic Monitoring and Management of Breast Cancer Patients' Symptoms
Brief Title: REBECCA - Research in Rehabilitation After Breast Cancer
Acronym: REBECCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: TRYG Foundation (Other); Rigshospitalet, Denmark (Other); Center for Kræft og Sundhed (Unknown)
Responsible Party: Principal Investigator, Christoffer Johansen, Professor, Head, Unit of Survivorship, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REBECCA
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Anxiety; Depression; Adverse Effects; Health Behavior
Keywords: neoplasms; rehabilitation; anxiety; depression; adverse effects; health behavior
MeSH Terms: conditions — Anxiety Disorders; Depression; Health Behavior; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening-based nurse navigation (Experimental): Based on systematic screening for psychological and physical symptoms as well as health behavior a nurse navigator will refer to and monitor use of appropriate rehabilitation programs
  Interventions: Other: Screening-based nurse navigation
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Screening-based nurse navigation — Screening-based nurse navigation for breast cancer rehabilitation
  Arms: Screening-based nurse navigation

SUMMARY:
The purpose of this study is to examine if a psychosocial intervention including a nurse navigator and systematic symptom screening may reduce psychological and physical symptoms as well as health behavior after breast cancer.

DETAILED DESCRIPTION:
In this pilot study with a randomized controlled trial design, we examine the effect of an intervention optimizing and integrating rehabilitation for breast cancer on psychological and physical symptoms as well as health behavior after breast cancer. In the intervention group, we systematically screen for psychological and physical symptoms as well as health behavior (smoking alcohol and physical activity) not in line with the recommendations. Patients who screen positive are offered a sequence of sessions with a navigator nurse who monitor rehabilitation needs, supports the patient, educate in self-management of symptoms and refer to existing rehabilitation services as well as to up to 6 free sessions with a psychologist specialized in cancer patients. The rehabilitation services that the nurse refers to include several hospital departments and municipality services as well as general practice and by thorough follow-up on the patients use of these, the intervention aims at developing an integrated treatment and rehabilitation trajectory. The control group receives standard care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary breast cancer at Breast Oncology Clinic, Rigshospitalet, Copenhagen, Denmark
* lives in Copenhagen municipality
* score ≥7 on distress thermometer
* able to read and understand Danish
* not pregnant
* expected survival more than 6 months
* physically able to participate in rehabilitation
* no severe psychiatric disease demanding treatment
* no severe cognitive problems (e.g. dementia or confusion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Psychological distress | 6 and 12 months
  Difference in change in psychological distress between patients in the intervention and control group.Psychological distress wil be measured using the Distress Thermometer

SECONDARY OUTCOMES:
Health related quality of life | 6 and 12 months
  Difference in change in patient reported health related quality of life between patients in the intervention and control group. Health related quality of life will be measured using the European Organization for Research and Treatment of Cancer quality of life questionnaire EORTC QLQ C30 and the EORTC BR23 including subscales.
Anxiety and depression | 6 and 12 months
  Difference in change in patient reported anxiety and depression between patients in the intervention and control group. Anxiety and depresison will be measured using the Hospital Anxiety and Depression scale (HADS).
Smoking | 6 and 12 months
  Difference in change in patient reported cigarette smoking measured in grams per day between patients in intervention and control group.
Alcohol consumption | 6 and 12 months
  Difference in change in patient reported alcohol consumption measured in grams per day between patients in intervention and control group.
Body mass index | 6 and 12 months
  Difference in change in patient reported body masss index between patients in intervention and control group.
Physical activity | 6 and 12 months
  Difference in change in patient reported physical activity between patients in intervention and control group.
Use of rehabilitation services | 6 and 12 months
  Difference in change in patient reported use of rehabilitation services between patients in intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, MD, Phd, Principal Investigator — Danish Cancer Society; Pernille E Bidstrup, MA. PhD, Principal Investigator — Danish Cancer Society
Locations (1):
- Rigshospitalet, Copenhagen, Denmark